CLINICAL TRIAL: NCT00956774
Title: Comparison of Three Cannulas for Hysterosalpingography: A Prospective, Randomized Study
Brief Title: Comparison of Three Cannulas for Hysterosalpingography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Comparison of 3 Cannulas - HSG
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2013-02

CONDITIONS: Infertility
Keywords: HSG; Cannula; HSG procedure; infertility evaluation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Balloon Catheter (Active Comparator)
  Interventions: Procedure: HSG with balloon catheter
- Cervical Vacuum Cup (Active Comparator)
  Interventions: Procedure: HSG with cervical vacuum cup
- acorn-tipped cannula (Active Comparator)
  Interventions: Procedure: HSG with acorn-tipped cannula

INTERVENTIONS:
Procedure: HSG with acorn-tipped cannula — Use of acorn-tipped cannula for HSG to evaluate tubal patency
  Arms: acorn-tipped cannula
Procedure: HSG with cervical vacuum cup — cup placed over cervix to create vacuum pressure.
  Arms: Cervical Vacuum Cup
Procedure: HSG with balloon catheter — balloon inserted via catheter into cervic for dilation.
  Arms: Balloon Catheter

SUMMARY:
The aim of this study is to compare the three commonly used hysterosalpingography (HSG) injection devices on the basis of patient pain perception, total fluoroscopic and procedural time, and side effects in a prospective, randomized study. An important and novel secondary outcome is the comparison of the quality of images obtained with these three devices. The investigators hypothesize that the balloon catheter and cervical vacuum cup will be less painful than the acorn tipped cannula and that there will be no difference in image quality between the three groups.

DETAILED DESCRIPTION:
This study is a prospective, randomized trial of women undergoing HSG as part of their infertility evaluation. At the time of scheduling, the patient will be randomized to either the cervical vacuum cup, balloon catheter (H/S catheter set, UA Medical, Biotech America), or the acorn-tipped cannula using stratified blocked randomization. 100 subjects will be randomized to one of the three cannulas. Patients will be stratified into 4 groups representative of the four reproductive endocrinologists in order to overcome any potential interoperator bias.

Four reproductive endocrinologists will perform the HSG procedures in a standardized fashion. Fluoroscopy will ensure proper location of the cannula and check for uterine filling of contrast. Digital images will document tubal filling and spilling of contrast. The patient will be rolled to right and left side to confirm free spillage of contrast in the peritoneal cavity. The last image will be taken after the balloon tip is deflated or the cannulas are removed to best evaluate the lower uterine segment.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing HSG at an academic medical center

Exclusion Criteria:

* Contrast media allergy
* Prior LEEP (Loop Electrosurgical Excision Procedure) or other cervical procedure
* Contraindication to NSAID use
* Known active pelvic infection
* Active vaginal bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
pain scores | 15 minutes

SECONDARY OUTCOMES:
the total duration of the procedure | 15 minutes
direct fluoroscopic time | 15 minutes
rates of vasovagal reaction | 15 minutes
diagnostic quality of images obtained | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Sara Lane, MD, Principal Investigator — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States